CLINICAL TRIAL: NCT06446141
Title: Effect of Osteopathic Technique on Respiratory Parameters and Pain in Thoracic Outlet Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Horus University (Other)
Responsible Party: Principal Investigator, Ahmed Metwally Mohamed Elshinnawy, Assistant Professor, Department of Physical Therapy for Neuromuscular Disorders and Its Surgery, Faculty of Physical Therapy, Horus University, New Damietta, Egypt, Horus University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HorusU1
Record Dates: First submitted 2024-06-01; First posted 2024-06-06 (Actual); Last update posted 2024-06-06 (Actual); Status verified 2024-06

CONDITIONS: Thoracic Outlet Syndrome
Keywords: Osteopathic Technique - Respiratory Parameters - Pain
MeSH Terms: conditions — Thoracic Outlet Syndrome

STUDY DESIGN:
Intervention Model Description: The Osteopathic technique included:
  Patients will be positioned in a supine position. Osteopathic technique will consist of supoccibital release, soft tissue release of thoracic outlet, mobilization of cervical facet joints, stretching of scalene anterior, scalene medius, upper trapezius, and levator scapula, pectorals major and minor. Subsequently, cost vertebral and cost transverse joint mobilizations will be applied using rib elevation. Then, manipulation of the vertebrae the levels between C6 and T1 will be applied using thrust mobilization technique. Afterwards, mobilization of the first rib will be applied. Finally, mobilization of the upper cervical spine will be performed.
Who Masked: Participant
Masking Description: I- Postural correction through correction of:
  * Forward head
  * Protracted shoulders
  * Depressed shoulder.
  II- Strengthen ex to:
  * Shoulder girdle elevators and retractors.
  * Cervical and dorsal extensors
  * raising arms to reach full flexion and elevation.
  III- Restoration of normal mobility
  o Inhibition of muscle spasm especially scaleni and pectoral ms. by source of heat& slow, sustain and self-stretching ex.
  IV- Breathing ex: diaphragmatic breathing.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): The Osteopathic technique included:
  Patients will be positioned in a supine position. Osteopathic technique will consist of supoccibital release, soft tissue release of thoracic outlet, mobilization of cervical facet joints, stretching of scalene anterior, scalene medius, upper trapezius, and levator scapula, pectorals major and minor. Subsequently, cost vertebral and cost transverse joint mobilizations will be applied using rib elevation. Then, manipulation of the vertebrae the levels between C6 and T1 will be applied using thrust mobilization technique. Afterwards, mobilization of the first rib will be applied. Finally, mobilization of the upper cervical spine will be performed.
  Interventions: Other: Osteopathic technique
- Group B (Active Comparator): I- Postural correction through correction of:
  * Forward head
  * Protracted shoulders
  * Depressed shoulder.
  II- Strengthen ex to:
  * Shoulder girdle elevators and retractors.
  * Cervical and dorsal extensors
  * raising arms to reach full flexion and elevation. III- Restoration of normal mobility o Inhibition of muscle spasm especially scaleni and pectoral ms. by source of heat& slow, sustain and self-stretching ex.
  IV- Breathing ex: diaphragmatic breathing,.
  Interventions: Other: Osteopathic technique

INTERVENTIONS:
Other: Osteopathic technique — Patients will be positioned in a supine position. Osteopathic technique will consist of supoccibital release, soft tissue release of thoracic outlet, mobilization of cervical facet joints, stretching of scalene anterior, scalene medius, upper trapezius, and levator scapula, pectorals major and minor. Subsequently, cost vertebral and cost transverse joint mobilizations will be applied using rib elevation. Then, manipulation of the vertebrae the levels between C6 and T1 will be applied using thrust mobilization technique. Afterwards, mobilization of the first rib will be applied. Finally, mobilization of the upper cervical spine will be performed.

SUMMARY:
Background: With regard to patients with thoracic outlet syndrome (GBS), it is important to improve inspiratory muscle strength and endurance, and pain perception in patients with TOS, so that patients are able to regain pulmonary function and endurance. Objective: To investigate the impact of osteopathic interventions on respiratory parameters and pain levels in individuals diagnosed with thoracic outlet syndrome (TOS). Subjects and methods: forty adults after the onset of TOS will be assigned randomly into two equal groups. In Group A will be allocated to traditional physical therapy program, three sessions/week in addition to 60-minute sessions of Osteopathic technique, one session/week for 3 months, group B will receive traditional physical therapy program, three sessions/week for 3 months. Selected respiratory parameters by spirometer, maximum inspiratory pressure (MIP) and maximum expiratory pressure (MEP) and a visual analogue scale of pain severity, measured at baseline and after 3 months.

DETAILED DESCRIPTION:
Method Design This parallel, two-group, randomized controlled trial will use concealed allocation, blinding of outcome assessors and intention-to- treat analysis. People with TOS will enroll to 3-month, osteopathic technique (Group A) or traditional physical therapy program (Group B). The allocation order will be concealed by placing each random allocation in a sealed opaque envelope, which will be opened after the participant enrolled in the study. Thus, researchers and therapists will not know or decide which enrolling participant would receive which therapy. After an envelope was opened, the participant and the therapists who administered the interventions will became aware of that participant's allocated intervention. Outcomes were measured at baseline and after 3 months. In addition to ethics approval ***********************.

Participants The study was conducted in Outpatient clinics of Faculty of physical therapy, Horus University. The study population will be consisted of patients diagnosed, by physicians or neurologists, as previous cases of 'deﬁnite' TOS. To be eligible to participate, patients with TOS were required to be aged 30-35 years, be in a stable clinical condition and have a physical disability based on assessment. The exclusion criteria were Patients with surgery plan for TOS, those who underwent TOS surgeries, those with smoking history, traumatic cervical injuries, diabetes mellitus and/or malignancies.

Measurement procedures:

1. Spirometer:
2. Micro Respiratory Pressure Meter:
3. Visual Analogue Scale:

Interventions Group A In addition to usual care from the treating physician or neurologist, participants will be prescribed a 3 months program. It will consist a 60 minute of traditional physical therapy program, three sessions/week in addition to 60-minute of Osteopathic technique, once per week.

The program included:

I- Postural correction through correction of:

* Forward head
* Protracted shoulders
* Depressed shoulder.

II- Strengthen ex to:

* Shoulder girdle elevators and retractors.
* Cervical and dorsal extensors
* raising arms to reach full flexion and elevation.

III- Restoration of normal mobility o Inhibition of muscle spasm especially scaleni and pectoral ms. by source of heat& slow, sustain and self-stretching ex.

IV- Breathing ex: diaphragmatic breathing.

The Osteopathic technique included:

Patients will be positioned in a supine position. Osteopathic technique will consist of supoccibital release, soft tissue release of thoracic outlet, mobilization of cervical facet joints, stretching of scalene anterior, scalene medius, upper trapezius, and levator scapula, pectorals major and minor. Subsequently, cost vertebral and cost transverse joint mobilizations will be applied using rib elevation. Then, manipulation of the vertebrae the levels between C6 and T1 will be applied using thrust mobilization technique. Afterwards, mobilization of the first rib will be applied. Finally, mobilization of the upper cervical spine will be performed.

Group B In addition to usual care from the treating physician or neurologist, participants were prescribed a 60 minute, three times per week of traditional physical therapy program.

The program included:

I- Postural correction through correction of:

* Forward head
* Protracted shoulders
* Depressed shoulder.

II- Strengthen ex to:

* Shoulder girdle elevators and retractors.
* Cervical and dorsal extensors
* raising arms to reach full flexion and elevation. III- Restoration of normal mobility o Inhibition of muscle spasm especially scaleni and pectoral ms. by source of heat& slow, sustain and self-stretching ex.

IV- Breathing ex: diaphragmatic breathing,.

ELIGIBILITY:
Inclusion Criteria:

* The study population consisted of patients diagnosed, by physicians or neurologists, as previous cases of 'deﬁnite' TOS.
* To be eligible to participate, patients with TOS were required to be aged 30-35 years, be in a stable clinical condition and have a physical disability based on assessment.

Exclusion Criteria:

* Patients with surgery plan for TOS, those who underwent TOS surgeries, those with smoking history, traumatic cervical injuries, diabetes mellitus and/or malignancies.

Ages: 30 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2024-05-01 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
(a) A portable spirometer: | 3 month
  (MIR Spirolab®) was used to measure pulmonary function test; forced vital capacity (FVC), forced expiratory volume in 1st second (FEV1), and Tiffeneau index (Forced expiratory volume in the one second/Forced vital capacity) (FEV1/FVC).
(b) Micro Respiratory Pressure Meter: | 3 month
  (MicroRPMTM made in USA). It was a handheld manometer with a disposal mouth-piece and used to calculate maximum inspiratory pressure (MIP) and maximum expiratory pressure (MEP)
(c) Visual Analogue Scale: | 3 month
  This scale was utilized to measure the pain intensity before and after treatment. The pain test was 10 cm (100 mm) length with two endpoints labeled (0=no pain) and (10=most pain ever).

CONTACTS AND LOCATIONS:
Overall Officials: Zeezy S. Eraky, Lecturer, Study Chair — Department of Physical Therapy for Internal Medicine and Elderly; Ehab A. Abdallah, Lecturer, Study Chair — Department of Orthopedic Physical Therapy; Haitham M. Elmasry, Lecturer, Study Chair — Department of Basic science; Hatem M. El-Samouly, Asst Prof, Study Chair — faculty of medicine
Locations (1):
- Horus University, Damietta, International Coastal Road New Damietta, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
All IPD will be shared through the corresponding author after acceptance of all authors